CLINICAL TRIAL: NCT03883386
Title: Loratadine for Improvement of Bone Pain in Patients With Chronic Granulocyte-Colony Stimulating Factor (G-CSF) Use
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Kelly Walkovich, Associate Professor of Pediatrics and Communicable Diseases, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HUM00152719
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Bone Pain
Keywords: Granulocyte-colony stimulating factor
MeSH Terms: interventions — Loratadine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Loratadine first (Experimental): Take treatment daily for 7 days.
  Interventions: Drug: Loratadine; Drug: Placebo
- Placebo first (Placebo Comparator): Take placebo daily for 7 days.
  Interventions: Drug: Loratadine; Drug: Placebo

INTERVENTIONS:
Drug: Loratadine — 10 mg in a capsule
  Other Names: Claritin
Drug: Placebo — Administered via capsule

SUMMARY:
G-CSF causes a release of histamine that may be a cause of chronic bone pain. Loratadine targets histamine, and so may be effective in reducing bone pain.The researchers plan to prospectively assess the effectiveness of loratadine for chronic bone pain in patients with chronic G-CSF use.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neutropenia
* Granulocyte-colony stimulating factor (G-CSF) use for at least 3 months at least 4 times per month
* Mean bone pain of at least a 2/10 as assessed by questions 3-6 of the Brief Pain Inventory (BPI)

Exclusion Criteria:

* Other sources of chronic pain
* Previously tried loratadine for 7 consecutive days or more for bone pain
* Allergy to loratadine
* Chronic daily usage of antihistamine without an acceptable alternative non-antihistamine medication

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Walkovich, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Assignment
Arm/Group | Loratadine First | Placebo First
Started | 2 | 1
Surveys Begun | 1 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Period: Washout and Second Assignment
Arm/Group | Loratadine First | Placebo First
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loratadine First | Placebo First | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 39 [22 to 55] | 60 [60 to 60] | 46 [22 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Severity Scores as Measured by the Brief Pain Inventory (BPI)
Description: The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning. The questions ask participants to rate their pain in the prior 24-hours OR prior 7-day on a 0 to 10 Numerical Rating Scale (NRS), where "0" indicates "No pain" and "10" indicates "Pain as bad as you can imagine."
  Modified BPI: Included the pain intensity subscale, it is a Numerical Rating Scale with 4 questions (3-6): each item is ranked where 0 is no pain - 10 the worst pain.
  The Modified BPI will be measured on Days 2, 4, and 6. The full BPI will be measured on Day 7. On day 7 only responses from questions 3-6 will be analyzed for this outcome and a mean composite score for Days 2, 4, 6, and 7 will be calculated.
Time Frame: Week 1 (baseline week), week 2 (placebo or loratadine), and week 4 (placebo or loratadine).
Population: Because only one participant completed an on-treatment survey, the data is not analyzable for any comparative purpose and therefore was not analyzed.
Groups:
- Loratadine: Take treatment daily for 7 days.
  Loratadine: 10 mg in a capsule
- Placebo: Take placebo by capsule daily for 7 days.
Arm/Group | Loratadine | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Pain Interference in Patients as Measured by the Brief Pain Inventory (BPI)
Description: Brief Pain Inventory (BPI) asks the participant to rate how their pain interferes with daily activities where "0" indicates "does not interfere and "10" indicates "completely interferes". The Pain Intensity Scale scores (Numerical Rating Scale (NRS)) for 7 questions: general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life from (BPI question 9A-G); 0 no life interference - 10 complete interference. Pain interference will be assessed on day 7 of each week.
Time Frame: Week 1 (baseline week), week 2 (placebo or loratadine), and week 4 (placebo or loratadine).
Population: as for outcome 1
Arm/Group | Loratadine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 weeks' following was planned; 2 weeks was the longest anyone actually participated.
Arm/Group | Loratadine First | Placebo First
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT03883386/Prot_SAP_000.pdf